CLINICAL TRIAL: NCT02608216
Title: [18F]Fluorothymidine (FLT) PET/CT Imaging in Rb+ Metastatic Breast Cancer Patients Undergoing LEE011 and Weekly Paclitaxel Therapy
Brief Title: [18F]FLT PET/CT in Rb+ Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 822997; NCT02774473 (obsolete NCT alias)
Record Dates: First submitted 2015-10-18; First posted 2015-11-18 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasm; Metastatic Breast Cancer; Rb+ Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — alovudine; Positron Emission Tomography Computed Tomography; ribociclib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FLT PET/CT (Experimental): All subjects will receive an [18F]FLT PET/CT scan.
  Interventions: Drug: [18F]FLT; Device: PET/CT; Drug: ribociclib; Drug: paclitaxel

INTERVENTIONS:
Drug: [18F]FLT — [18F]FLT PET/CT scan, imaging tracer
  Other Names: [18F]fluorothymidine
Device: PET/CT — [18F]FLT PET/CT scan
Drug: ribociclib — therapeutic
  Other Names: LEE011
Drug: paclitaxel — therapeutic

SUMMARY:
In this study positron emission tomography (PET/CT) imaging will be used to evaluate proliferative activity in sites of metastatic disease using the investigational radiotracer [18F]fluorothymidine (FLT).

DETAILED DESCRIPTION:
This protocol is designed to develop relationships between parameters determined from imaging biomarker studies and ones used for determination of therapeutic response to combined CDK4 Inhibitor and chemotherapy regimens. Imaging will occur prior to starting therapy on the separate therapeutic protocol UPCC 06115. Patients may undergo a second FLT PET/CT scan following a 3-day run of ribociclib (LEE011) (day -6 to -4) and a third FLT PET/CT scan on cycle 1 day 12 following two treatments of weekly Paclitaxel to compare changes in FLT uptake measures.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. History of histologically or cytologically confirmed breast cancer, any ER, PR or HER2 status is allowed as long as it expresses the Rb protein.
3. At least one site of metastatic breast cancer that is outside of the liver and bone that is identified by standard imaging (e.g. CT, MRI, FDG PET/CT, ultrasound, x-ray)
4. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.
5. Patients must be candidates to receive treatment on the therapeutic trial UPCC06115, a Phase I study of ribociclib (LEE011) and weekly paclitaxel.

Exclusion Criteria:

1. Females who are pregnant at the time of screening will not be eligible for this study, urine pregnancy test will be performed at screening in women of child-bearing potential.
2. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
3. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
4. Ineligible for the therapeutic trial UPCC 06115

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Measure changes in [18F]FLT uptake in metastatic tumors before and during treatment with ribociclib (LEE011) only, patient will have FLT PET/CT scan at baseline, run-in day -3, and cycle 1, day 1 of ribociclib (LEE011)/paclitaxel therapy | 4 years
  Measure changes in [18F]FLT uptake in metastatic tumors before and during treatment with ribociclib (LEE011) only and associate these changes with response to ribociclib (LEE011)/paclitaxel therapy.

SECONDARY OUTCOMES:
Measure changes in [18F]FLT uptake in metastatic tumors during and after treatment with ribociclib (LEE011) only, patient will have FLT PET/CT scan at baseline, run-in day -3, and cycle 1, day 1 of ribociclib (LEE011)/paclitaxel therapy | 4 years
  Measure changes in [18F]FLT uptake in metastatic tumors during and after treatment with ribociclib (LEE011) only and associate these changes with response to ribociclib (LEE011)/paclitaxel therapy.

CONTACTS AND LOCATIONS:
Overall Officials: David Mankoff, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Hospital, Philadelphia, Pennsylvania, United States